CLINICAL TRIAL: NCT02076828
Title: Comparison of Ferrous Sulfate, Polymaltose Complex and Iron-zinc in Iron Deficiency Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Yasemin Ozsurekci, Pediatric Infectious Diseases Specialist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HacettepeU
Record Dates: First submitted 2014-02-25; First posted 2014-03-04 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-02

CONDITIONS: Iron Deficiency Anemia
Keywords: anemia; iron polymaltose complexes; iron zinc
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fe-OH-PM (Santafer® sp.)(Group II) (Experimental): The patients in Group II were treated with Fe-OH-PM (Santafer® sp.), 6 mg/kg/day orally.
  Interventions: Drug: Santafer® sp.
- Fe-Zn (Ferro Zinc® sp.)(Group III) (Experimental): The patients in Group III were treated with Fe-Zn (Ferro Zinc® sp.), 6 mg/kg/day orally
  Interventions: Drug: Ferro Zinc® sp
- Fe-S (Ferro Sanol® sp.)(Group I) (Experimental): The patients in Group I were treated with Ferro Sanol® sp., 6 mg/kg/day orally
  Interventions: Drug: Ferro Sanol® sp

INTERVENTIONS:
Drug: Ferro Sanol® sp — The children with IDA that included in Fe-S (Ferro Sanol® sp.)(Group I) were treated with a therapeutic dose Ferro Sanol® sp as 6 mg/kg/day in the first 2 months and followed by maintenance treatment at a dosage of 2 mg/kg/day for the next 2 months.
  Other Names: Fe-S (Ferro Sanol® sp)(Group I)
  Arms: Fe-S (Ferro Sanol® sp.)(Group I)
Drug: Santafer® sp. — The children with IDA that included in Fe-OH-PM (Santafer® sp.)(Group II) were treated with a therapeutic dose Santafer® as 6 mg/kg/day in the first 2 months and followed by maintenance treatment at a dosage of 2 mg/kg/day for the next 2 months.
  Other Names: Fe-OH-PM (Santafer® sp.)(Group II)
  Arms: Fe-OH-PM (Santafer® sp.)(Group II)
Drug: Ferro Zinc® sp — The children with IDA that included in Fe-Zn (Ferro Zinc® sp.)(Group III) were treated with a therapeutic dose Ferro Zinc® sp. as 6 mg/kg/day in the first 2 months and followed by maintenance treatment at a dosage of 2 mg/kg/day for the next 2 months.
  Other Names: Fe-Zn (Ferro Zinc® sp.)(Group III)
  Arms: Fe-Zn (Ferro Zinc® sp.)(Group III)

SUMMARY:
The aim of the present study was to compare the effectiveness of the different oral iron preparations in children with IDA.

DETAILED DESCRIPTION:
Iron deficiency (ID) is the most common cause of the anemia throughout the world, with almost half of the population in developing countries suffering from ID. Children with iron deficiency anemia (IDA) may have functional consequences including impaired motor and physical growth. In the case of IDA, the underlying cause should be identified and treated. Iron supplementation remains an important strategy for the prevention and treatment of IDA and can produce substantial improvements in the functional performance of iron deficient individuals.

The iron-containing preparations available on the market vary widely in dosage, salt, and chemical state of iron (ferrous or ferric form). Current treatment strategy for IDA involves the oral use of Fe2+ salts (Fe SO4) and Fe3+ polymaltose complexes (FeOH3). Most of these preparations vary in their bioavailability, efficacy, side effects, and cost. Animal studies have not shown any significant difference in their oral bioavailability. However, in clinical practice, bivalent iron salts such as ferrous sulfate (Fe-S), ferrous gluconate, and ferrous fumarate are more widely used and are preferred over ferric iron preparations. Fe-S preparations usually present good bioavailability (between 10 and 15 %), while bioavailability of ferric iron preparations is 3 to 4 times less than that of conventional Fe-S. This is due to the extremely poor solubility of ferric iron in alkaline media and the fact that ferric iron needs to be transformed into ferrous iron before being absorbed. For this reason, among ferrous preparations, Fe-S remains the established and the standard treatment of ID due to its acceptable tolerability, high effectiveness, and low cost. The aim of the present study was to compare the effectiveness of the different oral iron preparations in children with IDA.

ELIGIBILITY:
Inclusion Criteria:

* The children with IDA, aged between 6 months and 15 years, were randomly included in Fe-S (Ferro Sanol® sp.)(Group I), Fe-OH-PM (Santafer® sp.)(Group II), and Fe-Zn (Ferro Zinc® sp.)(Group III). IDA was defined as hemoglobin (Hgb), serum iron and ferritin levels below -2SD according to age and gender.

Exclusion Criteria:

* The main exclusion criteria were anemia due to other causes except IDA
* Severe concurrent illness (cardiovascular, renal, and hepatic)
* Known hypersensitivity to ferrous or ferric preparations
* Malignancy of any type
* Children with thalassemia major, sickle cell anemia or other hemoglobinopathies, hemolytic anemia or aplastic or hypoplastic anemia.

Ages: 6 Months to 180 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Hb levels at 2 months | 2 months

SECONDARY OUTCOMES:
Change from baseline in Iron levels at 2 months. | 2 Months

OTHER OUTCOMES:
Improvements of the symptoms | 2 Months

CONTACTS AND LOCATIONS:
Overall Officials: Yasemin Ozsurekci, MD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Ankara/Sihhiye, Turkey (Türkiye)